CLINICAL TRIAL: NCT07053683
Title: Enhanced Efficacy of Early Orthopedic Intervention With Rapid Maxillary Expansion and Facemask Protraction on Skeletal and Quality of Life Outcomes in Class III Malocclusion: A Multicenter Randomized Controlled Trial
Brief Title: Efficacy of RME and Facemask Therapy for Class III Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Integrated Traditional Chinese and Western Medicine Hospital (Other)
Responsible Party: Principal Investigator, Lulu Wang, Principal investigator, Wuhan Integrated Traditional Chinese and Western Medicine Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WHH-ORTHO-2018-021
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Skeletal Class III Malocclusion
Keywords: Palatal Expansion Technique; Extraoral Traction Appliances; Malocclusion; Angle Class III; Cephalometry; Rapid Maxillary Expansion; Oral Health-Related Quality of Life
MeSH Terms: conditions — Malocclusion; Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: RME+FM Group (Experimental): Patients received a tooth-borne Hyrax-type rapid maxillary expander. After the active expansion phase, a Petit-type facemask was delivered, applying a forward and downward protraction force of 400-500g per side for 12-14 hours per day.
  Interventions: Device: Combined RME and Facemask Therapy
- Control: Facemask (FM) Alone Group (Active Comparator): Patients received the same facemask protraction therapy as the experimental group (same force, direction, and duration) but without undergoing RME. A removable mandibular occlusal splint was provided to disarticulate the occlusion.
  Interventions: Device: Facemask Therapy Alone

INTERVENTIONS:
Device: Combined RME and Facemask Therapy — This intervention involves two components. First, a tooth-borne Hyrax-type rapid maxillary expander is banded to the maxillary first permanent and deciduous molars. The screw is activated twice daily until posterior crossbite is overcorrected. Second, immediately following expansion, a Petit-type facemask is used to apply orthopedic protraction forces to the maxilla.
  Arms: Experimental: RME+FM Group
Device: Facemask Therapy Alone — This intervention involves the use of a Petit-type facemask to apply orthopedic protraction forces (400-500g per side, 12-14 hours/day) to the maxilla. A removable mandibular occlusal splint (flat bite plane) is used concurrently to facilitate anterior crossbite correction.
  Arms: Control: Facemask (FM) Alone Group

SUMMARY:
This multicenter randomized controlled trial compares the efficacy of Rapid Maxillary Expansion (RME) combined with facemask (FM) protraction versus FM protraction alone in treating growing children with skeletal Class III malocclusion. The study aims to evaluate the differences in vertical skeletal changes and Oral Health-Related Quality of Life (OHRQoL) between the two treatments.

DETAILED DESCRIPTION:
Skeletal Class III malocclusion is a challenging craniofacial anomaly, particularly prevalent in Asian populations. Early orthopedic intervention aims to correct the discrepancy and guide favorable growth. While facemask (FM) protraction is a standard treatment, its efficacy can be enhanced by Rapid Maxillary Expansion (RME), which is thought to disarticulate the circummaxillary sutures and facilitate a better orthopedic response. This prospective, multicenter, randomized controlled trial was designed to rigorously compare the combined RME+FM therapy against FM therapy alone. The study's primary objective was to assess the impact of these interventions on vertical skeletal dimensions, a key concern in Class III treatment. The secondary objective was to evaluate the patient-centered outcome of Oral Health-Related Quality of Life (OHRQoL). Eligible patients aged 7-12 were randomly assigned to one of two treatment groups. Cephalometric and OHRQoL data were collected at baseline and after 12 months of active treatment to determine if the combined approach offers superior clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal Class III malocclusion (ANB angle ≤ 0°) with a Wits appraisal ≤ -2 mm.
* Maxillary deficiency (SNA angle ≤ 80°).
* Prepubertal stage of skeletal development (Cervical Vertebral Maturation Stage CS1-CS3).
* Age between 7 and 12 years.
* Anterior crossbite or edge-to-edge incisor relationship.
* Angle Class III or end-on molar relationship.
* No previous orthodontic treatment.

Exclusion Criteria:

* Functional Class III malocclusion with no centric relation-centric occlusion discrepancy.
* Congenital craniofacial anomalies (e.g., cleft lip/palate).
* Severe systemic diseases.
* History of maxillofacial trauma.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 358 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Vertical Linear Cephalometric Measurements | Baseline, 12 Months
  Measured from standardized lateral cephalograms and Cone-Beam Computed Tomography (CBCT) scans. Key measurements include overbite (mm), maxillary molar vertical position (PP-Ms distance, mm), and maxillary anterior position (X-A distance, mm).
Change in Angular Cephalometric Measurements | Baseline, 12 Months
  Measured from standardized lateral cephalograms and CBCT scans. Key measurements include sagittal jaw relationship (ANB angle, degrees), mandibular plane angle (SN-MP, degrees), and palatal plane angle (SN-PP, degrees).

SECONDARY OUTCOMES:
Change in Dental Positional Measurements | Baseline (T0) and 6-month follow-up (T1).
  Change in cephalometric measurements assessing the position and inclination of the incisors, including the UI-NA angle, UI-LI angle (upper to lower incisor angle), UI-NA distance (upper incisor protrusion), and LI-NB distance (lower incisor position). These are measured in degrees or millimeters as appropriate.
Change in Dental Cephalometric Measurements | Baseline, 12 Months
  Measured from lateral cephalograms to assess changes in the inclination of the maxillary and mandibular incisors.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan No.1 Hospital, Wuhan, Hubei, China